CLINICAL TRIAL: NCT01736202
Title: Acute Effects of an Oral Fat Load on Skeletal Muscle and Hepatic Insulin Sensitivity (FLAME-study)
Brief Title: Acute Effects of an Oral Fat Load on Skeletal Muscle and Hepatic Insulin Sensitivity
Acronym: FLAME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: German Diabetes Center (Other)
Collaborators: German Center for Diabetes Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: FLAME
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Last update posted 2023-08-25 (Actual); Status verified 2023-06

CONDITIONS: Insulin Sensitivity
Keywords: oral fat; insulin sensitivity
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Palm oil orally (Active Comparator): oral fat load
  Interventions: Biological: fat orally
- Canola oil orally (Active Comparator): Oral fat load
  Interventions: Biological: fat orally
- Water orally (Placebo Comparator): oral water administration as control
  Interventions: Biological: fat orally

INTERVENTIONS:
Biological: fat orally — Oral ingestion of palm oil or canola oil or water at timepoint zero
  Other Names: water orally

SUMMARY:
The development of type 2 diabetes is based on a combination of insulin resistance and beta cell dysfunction. In the last years, elevated FFA were recognized as a key players in the pathogenesis of insulin resistance and type 2 diabetes.

The study compares the acute effects of an oral lipid bolus on insulin sensitivity and hepatic glucose metabolism in healthy humans.

DETAILED DESCRIPTION:
A dysregulation of lipid metabolism with increased levels of free fatty acids (FFA) represents one key mechanism in the pathogenesis of insulin resistance, which contributes to the development of type 2 diabetes (T2D). In most cases, dyslipidemia is related to obesity and the metabolic syndrome. Not only skeletal muscle glucose uptake, but also hepatic glucose fluxes are altered in insulin resistant states. In obese and T2D subjects, rates of gluconeogenesis (GNG) are increased, but in obese normoglycemic subjects endogenous glucose production (EGP) remains constant because of downregulation of glycogenolysis (GL). However, in T2D subjects, both GNG and GL are elevated, contributing to fasting and postprandial hyperglycemia. Therefore, elevated GNG rates may represent an early event in the pathophysiology of insulin resistance and T2D.

Preliminary studies of our institute show that intravenous lipid infusion with subsequent elevation of FFA results in increased GNG rates without alteration of EGP in lean, non-diabetic subjects. In another recent study we investigated the effects of an oral fat load on hepatic insulin sensitivity. As expected, we did not find any alterations in EGP; however, rates of GNG and GL have not been assessed.

The aim of this study is to analyze the effects of an oral fat load with transiently elevated levels of circulating lipids on hepatic glucose fluxes, especially GNG and GL, to elucidate the role of dietary fat in the induction of insulin resistance in healthy humans.

In this randomized, controlled cross-over study, effects of oral palm oil and canola oil ingestion will be investigated in young, healthy lean subjects. Hepatic glucose fluxes will be assessed by two independent methods, in vivo magnet resonance spectroscopy (MRS) and the deuterated water/acetaminophen method, which also allows for the determination of glycogen cycling rates. Furthermore, hepatic phosphorus metabolites and liver fat content will be monitored by MRS.

ELIGIBILITY:
Inclusion Criteria:

* healthy male and female subjects
* age 20-40
* BMI 20-25 kg/m2

Exclusion Criteria:

* hyperlipidemia
* smoking
* pregnancy
* allergy against paracetamol/palm oil/canola oil
* contraindication for MRI investigations
* anaemia
* taking drugs influencing lipid or glucose metabolism, the immune system or antihypertensive treatment
* M. Meulengracht
* Hepatitis/HIV
* chronic diseases

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03; Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Change in rate of glucose disappearance (Rd) | 6 hours
  Measurement of whole body insulin sensitivity in a hyperinsulinamic euglicamic clamp with deuterated glucose kinetics

SECONDARY OUTCOMES:
Change in rate of hepatic endogenous glucose production (EGP) | 6 hours
  Measurement of hepatic EGP in a hyperinsulinamic euglicamic clamp with deuterated glucose kinetics

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, Prof., MD, Study Director — German Diabetes Center
Locations (1):
- German Diabetes Center, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Sarabhai T, Koliaki C, Mastrototaro L, Kahl S, Pesta D, Apostolopoulou M, Wolkersdorfer M, Bonner AC, Bobrov P, Markgraf DF, Herder C, Roden M. Dietary palmitate and oleate differently modulate insulin sensitivity in human skeletal muscle. Diabetologia. 2022 Feb;65(2):301-314. doi: 10.1007/s00125-021-05596-z. Epub 2021 Oct 26. PMID 34704121
- [Derived] Sarabhai T, Kahl S, Szendroedi J, Markgraf DF, Zaharia OP, Barosa C, Herder C, Wickrath F, Bobrov P, Hwang JH, Jones JG, Roden M. Monounsaturated fat rapidly induces hepatic gluconeogenesis and whole-body insulin resistance. JCI Insight. 2020 May 21;5(10):e134520. doi: 10.1172/jci.insight.134520. PMID 32434996
- [Derived] Hernandez EA, Kahl S, Seelig A, Begovatz P, Irmler M, Kupriyanova Y, Nowotny B, Nowotny P, Herder C, Barosa C, Carvalho F, Rozman J, Neschen S, Jones JG, Beckers J, de Angelis MH, Roden M. Acute dietary fat intake initiates alterations in energy metabolism and insulin resistance. J Clin Invest. 2017 Feb 1;127(2):695-708. doi: 10.1172/JCI89444. Epub 2017 Jan 23. PMID 28112681